CLINICAL TRIAL: NCT02577042
Title: Study of the Effect of Atorvastatin for Reducing "Inflaming" (Aging-related Complication) in HIV-infected Patients Older Than 45 Years Receiving a Protease Inhibitor-based Regimen Versus a Raltegravir-based Regimen
Brief Title: Study of the Effect of Atorvastatin for Reducing Aging-related Complication in HIV-infected Patients Older Than 45 Years Receiving a Protease Inhibitor-based Regimen Versus a Raltegravir-based Regimen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RALATOR
Record Dates: First submitted 2015-10-07; First posted 2015-10-16 (Estimated); Results first posted 2020-06-22 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Aging-related Inflammation in HIV-infected Patients
Keywords: Raltegravir; protease inhibitors; darunavir; inflammation; statins; comorbidities
MeSH Terms: conditions — Inflammation | interventions — Raltegravir Potassium; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Raltegravir + Atorvastatin (Experimental): Switching the PI by raltegravir, plus Kivexa or Truvada, for 24 weeks. After that, atorvastatin, 20mg/day, will be added for 48 weeks
  Interventions: Drug: Raltegravir; Drug: Atorvastatin
- PI-based regimen + Atorvastatin (Active Comparator): Continue with the same PI-based regimen, plus Kivexa or Truvada, for 24 weeks. After that, atorvastatin, 20mg/day, will be added for 48 weeks.
  Interventions: Drug: PI-based regimen; Drug: Atorvastatin

INTERVENTIONS:
Drug: Raltegravir — Switching the PI by raltegravir 400mg every 12 hours, plus Kivexa or Truvada, for 24 weeks.
  Arms: Raltegravir + Atorvastatin
Drug: PI-based regimen — Continue with the same PI-based regimen, plus Kivexa or Truvada, for 24 weeks.
  Arms: PI-based regimen + Atorvastatin
Drug: Atorvastatin — Atorvastatin, 20mg/day, will be added after 24 weeks of study for 48 weeks

SUMMARY:
Physicians in charge of HIV-infected patients are increasingly being faced to previously unrecognized comorbid conditions such as atherosclerosis and cardiovascular events, loss of renal function, osteopenia/osteoporosis and bone fractures or non-AIDS-defining cancers (1-4). The incidence of these conditions seems to be higher than in the general population but there are controversial data about if these diseases appear at a younger age in HIV-infected patients.

The investigators propose a strategy for treatment of elderly HIV-infected patients with a double impact on systemic inflammation and age-related co-morbidities by switching the protease inhibitors by raltegravir, a integrase inhibitor with a neutral effect on lipid and bone metabolism, and adding an statin because of their anti-inflammatory effect. For safety reasons, only patients with maintained viral suppression (documented indetectable viral load for 1 year or more), and no history of virological failure to integrase inhibitors or suspected or documented resistance mutations to the integrase or retrotranscriptase will be candidates for the study.

Interleukin -6 and D-dimer are biomarkers that most strongly predict mortality in treated HIV infection and sCD14, sCD163 are soluble markers of monocyte activation that reflect a key source of inflammation and coagulation in HIV infection and predict mortality (26,27). For that reasons, these markers were chosen to determine changes on them after the introduction of the statin and the change of antiretrovirals

DETAILED DESCRIPTION:
Physicians in charge of HIV-infected patients are increasingly being faced to previously unrecognized comorbid conditions such as atherosclerosis and cardiovascular events, loss of renal function, osteopenia/osteoporosis and bone fractures or non-AIDS-defining cancers (1-4).

The incidence of these conditions seems to be higher than in the general population but there are controversial data about if these diseases appear at a younger age in HIV-infected patients.

Different pathogenic mechanisms are involved in the increased risk of comorbidities. First, the increased life expectancy of the HIV-infected population. The number of elderly HIV+ individuals is dramatically increasing, and nowadays, approximately one-half of the people living with HIV in the United States are age 50 or older (5). In this sense, aging itself is a condition associated with a chronic inflammation and immune senescence, contributing to accelerate age-related morbidity. Second, the persistent inflammatory state and activation of the immune system also induced by the HIV-infection, per se. This condition amplifies the risk of age-related morbidity (6-9). Finally, antiretroviral-related toxicities contribute to accelerate the apparition of some of these diseases such as the dyslipidemia and cardiovascular events (mainly associated with the protease inhibitors use), renal damage or low bone mineral density (especially by tenofovir and probably also by protease inhibitors).

As a consequence, one of the current aims of HIV management is the management of chronic non-infectious co-morbidities in an increasingly older and more complex population. The use of the newest and more safety antiretroviral drugs is a mandatory strategy, especially in this elderly population, to achieve a maintained viral suppression. However, there are many published studies showing higher levels of inflammation even in patients under a viral suppression, in comparison with general population. Regarding this condition, the investigators currently lack effective interventions to potently block this inflammatory status. Although some initial data are published about this regard, data in elderly HIV-infected people are lacking.

Based on these data, the investigators propose a strategy for treatment of elderly HIV-infected patients with a double impact on systemic inflammation and age-related co-morbidities by switching the protease inhibitors by raltegravir, a integrase inhibitor with a neutral effect on lipid and bone metabolism, and adding an statin because of their anti-inflammatory effect. For safety reasons, only patients with maintained viral suppression (documented indetectable viral load for 1 year or more), and no history of virological failure to integrase inhibitors or suspected or documented resistance mutations to the integrase or retrotranscription will be candidates for the study.

Raltegravir is an antiretroviral drug that received approval by the U.S. Food and Drug Administration (FDA) in 2007. It was the first of a new class of HIV drugs, the integrase inhibitors, and exhibited rapid, potent and durable antiretroviral activity in antiretroviral naïve patients and in treatment-experienced patients with drug-resistant HIV-1 (10-12). Raltegravir has demonstrated a neutral effect on lipid and renal parameters, and a better impact on bone mineral density (13) and lipid profile than protease inhibitors (14).

Statins are lipid-lowering drugs that also exert anti-inflammatory effects, and have immune-modulatory properties. Recent studies in HIV-infected population have suggested that statins have an anti-inflammatory effect, evaluated by inflammatory markers (15-21), and that the statin use is associated with a lower risk of non-AIDS defining morbidities and malignancies and mortality (22-25). But limited data have been published, mainly based on retrospective studies, and no clinical recommendations are available. The investigators propose the use of atorvastatin to study the anti-inflammatory effect measuring changes in inflammatory markers and some clinical conditions. Atorvastatin was chosen due to the low drug-drug interactions of this statin and ritonavir and the low cost. Since very few data are available about the effect of statins on inflammatory markers and clinical conditions, a intermediate dose (20 mg per day) was selected.

IL-6 and D-dimer are biomarkers that most strongly predict mortality in treated HIV infection and sCD14, sCD163 are soluble markers of monocyte activation that reflect a key source of inflammation and coagulation in HIV infection and predict mortality (26,27). For that reasons, these markers were chosen to determine changes on them after the introduction of the statin and the change of antiretrovirals.

ELIGIBILITY:
Inclusion Criteria:

* Patient having a diagnosis of HIV-1 infection.
* Age 45 years old.
* Current highly active antiretroviral therapy including Truvada or Kivexa plus a ritonavir boosted PI started at least 3 months before.
* Maintained undetectable plasma HIV-1 RNA (VL < 50 copies/mL) for at least 12 months.
* Voluntary written informed consent.

Exclusion Criteria:

* History of virological failure to integrase inhibitors.
* Suspected or documented resistance mutations to the integrase, as well as NRTI-related mutations that may impact nucleoside activity in current regimen.
* Systemic concurrent process such as coinfection with hepatitis C or B, acute systemic infection within the last 4 months, neoplasm, chronic inflammatory process, etc.
* Treatment with other drugs with anti-inflammatory, anticoagulant or antiplatelet effect (for instance corticosteroids, aspirin, etc…)
* Therapy with statins within the last 6 months.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain

REFERENCES:
- [Derived] Negredo E, Jimenez M, Puig J, Loste C, Perez-Alvarez N, Urrea V, Echeverria P, Bonjoch A, Clotet B, Blanco J. A randomized pilot trial to evaluate the benefit of the concomitant use of atorvastatin and Raltegravir on immunological markers in protease-inhibitor-treated subjects living with HIV. PLoS One. 2020 Sep 17;15(9):e0238575. doi: 10.1371/journal.pone.0238575. eCollection 2020. PMID 32941476
- [Derived] Negredo E, Estrada V, Domingo P, Gutierrez MD, Mateo GM, Puig J, Bonjoch A, Ornelas A, Echeverria P, Estany C, Toro J, Clotet B. Switching from a ritonavir-boosted PI to dolutegravir as an alternative strategy in virologically suppressed HIV-infected individuals. J Antimicrob Chemother. 2017 Mar 1;72(3):844-849. doi: 10.1093/jac/dkw504. PMID 27999056

RESULTS

PARTICIPANT FLOW:
Groups:
- Raltegravir + Atorvastatin: Switching the PI by raltegravir, plus Kivexaâ or Truvada, for 24 weeks. After that, atorvastatin, 20mg/day, will be added for 48 weeks
  Raltegravir: Switching the PI by raltegravir 400mg every 12 hours, plus Kivexa or Truvada, for 24 weeks.
  Atorvastatin: Atorvastatin, 20mg/day, will be added after 24 weeks of study for 48 weeks
Period: Overall Study
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Started | 20 | 22
Completed | 15 | 19
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 22 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 49.5 (3.5) | 51.8 (8.2) | 50.65 (5.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 18 | 17 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 22 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Inflammatory Marker IL-6
Description: Switching the PI by raltegravir, plus Kivexa or Truvada for 24 weeks. After that, atorvastatin, 20mg/day has been added for 48 weeks. (intergroup and intragroup)
Time Frame: baseline, wk24 and wk72
Measure: Mean (Inter-Quartile Range); unit: pg/mL
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 20 | 22
pg/mL
  Baseline | 42.5 [34.5 to 50.1] | 40.0 [36.9 to 53.7]
  week 24 | 39.3 [34.6 to 49.8] | 41.1 [36.1 to 53.2]
  week 72 | 43.2 [36.8 to 52.9] | 41.7 [34.7 to 51.5]

2. Primary Outcome: Changes in Plasma Soluble Markers (D-dimer)
Description: Changes in plasma soluble markers (D-dimer)
Time Frame: baseline, wk24 and wk72
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 20 | 22
ng/mL
  Baseline | 1743 [1459 to 1894] | 1990 [1574 to 2523]
  wk24 | 1844 [1547 to 2340] | 1917 [1552 to 2244]
  wk72 | 2051 [1656 to 2414] | 1868 [1438 to 2175]

3. Other Pre Specified Outcome: Changes in the Inflammatory, Immune and Coagulation
Description: Changes in the inflammatory, immune and coagulation (intergroup and intragroup )
Time Frame: at week 72 from week 24 to assess the effect of statin
Population: Data were not collected
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Compare Intergroup and Intragroup Changes in the Inflammatory, Immune and Coagulation
Description: Compare intergroup and intragroup changes in the inflammatory, immune and coagulation
Time Frame: at week 72 from baseline to assess the effect of PI or raltegravir plus statin
Population: Data were not collected
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Compare Intergroup and Intragroup Changes in the Inflammatory, Immune and Coagulation
Description: Compare intergroup and intragroup changes in the inflammatory, immune and coagulation
Time Frame: at week 24 from baseline to asses the effect of PI or raltegravir
Population: Data were not collected
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Compare Intergroup and Intragroup Changes in Lipid Profile
Description: Compare intergroup and intragroup changes in lipid profile
Time Frame: at week 72 from week 24 to assess the effect of statin
Population: Data were not collected
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Compare Intergroup and Intragroup Changes in Lipid Profile
Description: Compare intergroup and intragroup changes in lipid profile
Time Frame: at week 72 from baseline to assess the effect of PI or raltegravir plus statin
Population: Data were not collected
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Compare Intergroup and Intragroup Changes in Lipid Profile
Description: Compare intergroup and intragroup changes in lipid profile
Time Frame: at week 24 from baseline to asses the effect of PI or raltegravir
Population: Data were not collected
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Compare Intergroup and Intragroup Changes in Lumbar and Femoral BMD and T-score Measured by DEXA
Description: Compare intergroup and intragroup changes in lumbar and femoral BMD and t-score measured by DEXA
Time Frame: at week 72 from week 24 to assess the effect of statin
Population: Data were not collected
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Compare Intergroup and Intragroup Changes in Lumbar and Femoral BMD and T-score Measured by DEXA
Description: Compare intergroup and intragroup changes in lumbar and femoral BMD and t-score measured by DEXA
Time Frame: at week 72 from baseline to assess the effect of PI or raltegravir plus statin
Population: Data were not collected
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Compare Intergroup and Intragroup Changes in Lumbar and Femoral BMD and T-score Measured by DEXA
Description: Compare intergroup and intragroup changes in lumbar and femoral BMD and t-score measured by DEXA
Time Frame: at week 24 from baseline to asses the effect of PI or raltegravir
Population: Data were not collected
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Compare Intergroup and Intragroup Changes in Bone Turnover Markers
Description: Compare intergroup and intragroup changes in bone turnover markers
Time Frame: at week 72 from week 24 to assess the effect of statin
Population: Data were not collected
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Compare Intergroup and Intragroup Changes in Bone Turnover Markers
Description: Compare intergroup and intragroup changes in bone turnover markers
Time Frame: at week 72 from baseline to assess the effect of PI or raltegravir plus statin
Population: Data were not collected
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: Compare Intergroup and Intragroup Changes in Bone Turnover Markers
Description: Compare intergroup and intragroup changes in bone turnover markers
Time Frame: at week 24 from baseline to asses the effect of PI or raltegravir
Population: Data were not collected
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 0 | 0

15. Other Pre Specified Outcome: Compare Intergroup and Intragroup Changes in Renal Parameters
Description: Compare intergroup and intragroup changes in renal parameters
Time Frame: at week 72 from week 24 to assess the effect of statin
Population: Data were not collected
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 0 | 0

16. Other Pre Specified Outcome: Compare Intergroup and Intragroup Changes in Renal Parameters
Description: Compare intergroup and intragroup changes in renal parameters
Time Frame: at week 72 from baseline to assess the effect of PI or raltegravir plus statin
Population: Data were not collected
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 0 | 0

17. Other Pre Specified Outcome: Compare Intergroup and Intragroup Changes in Renal Parameters
Description: Compare intergroup and intragroup changes in renal parameters
Time Frame: at week 24 from baseline to asses the effect of PI or raltegravir
Population: Data were not collected
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 0 | 0

18. Other Pre Specified Outcome: Viral Load < 50 Copies
Description: viral load < 50 copies
Time Frame: at week 72
Population: Data were not collected
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 0 | 0

19. Other Pre Specified Outcome: Viral Load > 50 Copies
Description: viral load > 50 copies
Time Frame: through study completion
Population: Data were not collected
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 0 | 0

20. Other Pre Specified Outcome: CD4+/CD8+ T Lymphocytes
Description: CD4+/CD8+ T lymphocytes
Time Frame: at week 72 from baseline
Population: Data were not collected
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline to week 72
Arm/Group | Raltegravir + Atorvastatin | PI-based Regimen + Atorvastatin
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 3/20 | 0/22
Other Adverse Events (participants affected / at risk) | 0/20 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Raltegravir + Atorvastatin (N=20) | PI-based Regimen + Atorvastatin (N=22)
increments of creatine kinase (Cardiac disorders) | 2 | 0
increment of liver enzymes (Hepatobiliary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT02577042/Prot_SAP_000.pdf